CLINICAL TRIAL: NCT03937219
Title: A Randomized, Double-Blind, Controlled Phase 3 Study of Cabozantinib in Combination With Nivolumab and Ipilimumab Versus Nivolumab and Ipilimumab in Subjects With Previously Untreated Advanced or Metastatic Renal Cell Carcinoma of Intermediate or Poor Risk
Brief Title: Study of Cabozantinib in Combination With Nivolumab and Ipilimumab in Patients With Previously Untreated Advanced or Metastatic Renal Cell Carcinoma
Acronym: COSMIC-313
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XL184-313; 2024-515616-47-00 (EU CTIS Number)
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Renal Cell Carcinoma
Keywords: renal; cancer; carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms; Carcinoma | interventions — cabozantinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Approximately 840 eligible subjects with intermediate- or poor-risk advanced or metastatic RCC by IMDC criteria will be randomized in a 1:1 ratio.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Cabozantinib + nivolumab + ipilimumab (4 doses) followed by cabozantinib + nivolumab
  Interventions: Drug: Cabozantinib; Biological: Nivolumab; Biological: Ipilimumab
- Control Arm (Active Comparator): Cabozantinib-matched placebo + nivolumab + ipilimumab (4 doses) followed by cabozantinib-matched placebo + nivolumab
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Drug: Cabozantinib-matched placebo

INTERVENTIONS:
Drug: Cabozantinib — Specified dose on specified days.
  Other Names: Cabometyx; XL184
  Arms: Experimental Arm
Biological: Nivolumab — Specified dose on specified days.
  Other Names: Opdivo; BMS-936558
Biological: Ipilimumab — Specified dose on specified days.
  Other Names: Yervoy; BMS-734016
Drug: Cabozantinib-matched placebo — Specified dose on specified days.
  Arms: Control Arm

SUMMARY:
This is a multicenter, randomized, double-blinded, controlled Phase 3 trial of cabozantinib in combination with nivolumab and ipilimumab versus nivolumab and ipilimumab in combination with matched placebo. Approximately 840 eligible subjects with intermediate- or poor-risk advanced or metastatic RCC by IMDC criteria will be randomized in a 1:1 ratio at approximately 180 sites.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, controlled Phase 3 trial of cabozantinib in combination with nivolumab and ipilimumab versus nivolumab and ipilimumab in combination with matched placebo. The primary objective of this study is to evaluate the effect of cabozantinib in combination with nivolumab and ipilimumab ("triplet") on the duration of progression-free survival (PFS) versus nivolumab and ipilimumab. A secondary objective is to evaluate the effect of triplet combination on the duration of overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) renal cell carcinoma with a clear-cell component.
* Intermediate- or poor-risk RCC as defined by International Metastatic RCC Database Consortium (IMDC) criteria.
* Measurable disease per RECIST 1.1 as determined by the Investigator. Measurable disease must be outside the radiation field if radiation therapy was previously administered.
* Karnofsky Performance Status (KPS) ≥ 70%.
* Adequate organ and marrow function.

Exclusion Criteria:

* Prior systemic anticancer therapy for unresectable locally advanced or metastatic RCC including investigational agents.
* Radiation therapy for bone metastasis within 2 weeks, any other radiation therapy within 4 weeks prior to randomization.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and stable for at least 4 weeks prior to randomization.
* Concomitant anticoagulation with oral anticoagulants or platelet inhibitors.
* Administration of a live, attenuated vaccine within 30 days prior to randomization.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to serious cardiovascular disorders (including uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment), GI disorders associated with high risk for perforation or fistula formation, tumors invading GI tract, bowel obstruction, intra-abdominal abscess, clinically significant bleeding events, cavitating pulmonary lesions, or lesions invading major pulmonary blood vessels.
* Other clinically significant disorders such as:

  * Autoimmune disease that has been symptomatic or required treatment within the past two years from the date of randomization.
  * Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization.
  * Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active myobacterial infection.
  * Known history of COVID-19 unless the subject has clinically recovered from the disease at least 30 days prior to randomization.
* Major surgery (eg, nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 4 weeks prior to randomization. Minor surgeries within 10 days prior to randomization. Subjects must have complete wound healing from major or minor surgery before randomization.
* Any other active malignancy at time of randomization or diagnosis of another malignancy within 3 years prior to randomization that requires active treatment, except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2027-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (159):
- United States (30):
  - Exelixis Clinical Site #116, La Jolla, California
  - Exelixis Clinical Site #166, Orange, California
  - Exelixis Clinical Site #29, Boca Raton, Florida
  - Exelixis Clinical Site #44, Miami, Florida
  - Exelixis Clinical Site #3, Atlanta, Georgia
  - Exelixis Clinical Site #95, Chicago, Illinois
  - Exelixis Clinical Site #69, Scarborough, Maine
  - Exelixis Clinical Site #58A, Baltimore, Maryland
  - Exelixis Clinical Site #7B, Boston, Massachusetts
  - Exelixis Clinical Site #7A, Boston, Massachusetts
  - Exelixis Clinical Site #7C, Boston, Massachusetts
  - Exelixis Clinical Site #6, Burlington, Massachusetts
  - Exelixis Clinical Site #15, Detroit, Michigan
  - Exelixis Clinical Site #24, Kansas City, Missouri
  - Exelixis Clinical Site #4, St Louis, Missouri
  - Exelixis Clinical Site #2, Omaha, Nebraska
  - Exelixis Clinical Site #159, New York, New York
  - Exelixis Clinical Site #8, New York, New York
  - Exelixis Clinical Site #19, Syracuse, New York
  - Exelixis Clinical Site #101, Charlotte, North Carolina
  - Exelixis Clinical Site #107, Portland, Oregon
  - Exelixis Clinical Site #12, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #102, Charleston, South Carolina
  - Exelixis Clinical Site #5, Myrtle Beach, South Carolina
  - Exelixis Clinical Site #10, Nashville, Tennessee
  - Exelixis Clinical Site #38, Nashville, Tennessee
  - Exelixis Clinical Site #64, Fairfax, Virginia
  - Exelixis Clinical Site #57, Seattle, Washington
  - Exelixis Clinical Site #1, Spokane, Washington
  - Exelixis Clinical Site #13, Madison, Wisconsin
- Argentina (7):
  - Exelixis Clinical Site #153, Pilar, Buenos Aires
  - Exelixis Clinical Site #109, Rosario, Santa Fe Province
  - Exelixis Clinical Site #73, San Miguel de Tucumán, Tucumán Province
  - Exelixis Clinical Site #54, Buenos Aires
  - Exelixis Clinical Site #63, CABA
  - Exelixis Clinical Site #110, Ciudad Autonoma de Buenos Aire
  - Exelixis Clinical Site #120, Córdoba
- Australia (11):
  - Exelixis Clinical Site #32, Albury, New South Wales
  - Exelixis Clinical Site #35, Kogarah, New South Wales
  - Exelixis Clinical Site #27, North Ryde, New South Wales
  - Exelixis Clinical Site #33, Sydney, New South Wales
  - Exelixis Clinical Site #17, South Brisbane, Queensland
  - Exelixis Clinical Site #14, Woolloongabba, Queensland
  - Exelixis Clinical Site #18, Adelaide, South Australia
  - Exelixis Clinical Site #11, North Adelaide, South Australia
  - Exelixis Clinical Site #9, Ballarat, Victoria
  - Exelixis Clinical Site #23, Box Hill, Victoria
  - Exelixis Clinical Site #26, Subiaco, Western Australia
- Austria (4):
  - Exelixis Clinical Site #98, Wiener Neustadt, Lower Austria
  - Exelixis Clinical Site #76, Linz, Upper Austria
  - Exelixis Clinical Site #75, Salzburg
  - Exelixis Clinical Site #126, Vienna
- Belgium (2):
  - Exelixis Clinical Site #112, Brussels
  - Exelixis Clinical Site #146, Hasselt
- Brazil (9):
  - Exelixis Clinical Site #154, Belo Horizonte, Minas Gerais
  - Exelixis Clinical Site #155, Curitiba, Paraná
  - Exelixis Clinical Site #158, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #140, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #163, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #168, Barretos, São Paulo
  - Exelixis Clinical Site #162, São José do Rio Preto, São Paulo
  - Exelixis Clinical Site #119, São Paulo
  - Exelixis Clinical Site #141, São Paulo
- Canada (5):
  - Exelixis Clinical Site #22, Calgary, Alberta
  - Exelixis Clinical Site #105, Winnipeg, Manitoba
  - Exelixis Clinical Site #46, Ottawa, Ontario
  - Exelixis Clinical Site #25, Toronto, Ontario
  - Exelixis Clinical Site #113, Montreal, Quebec
- Chile (3):
  - Exelixis Clinical Site #85, Temuco, Región de La Araucanía (IX)
  - Exelixis Clinical Site #91, Santiago
  - Exelixis Clinical Site #100, Santiago
- Czechia (3):
  - Exelixis Clinical Site #89, Králová
  - Exelixis Clinical Site #114, Prague
  - Exelixis Clinical Site #118, Prague
- Finland (3):
  - Exelixis Clinical Site #50, Helsinki
  - Exelixis Clinical Site #56, Tampere
  - Exelixis Clinical Site #52, Turku
- France (13):
  - Exelixis Clinical Site #86, Bordeaux
  - Exelixis Clinical Site #71, Le Mans
  - Exelixis Clinical Site #78, Lyon
  - Exelixis Clinical Site #80, Montpellier
  - Exelixis Clinical Site #66, Nice
  - Exelixis Clinical Site #150, Paris
  - Exelixis Clinical Site #65, Reims
  - Exelixis Clinical Site #125, Rennes
  - Exelixis Clinical Site #128, Strasbourg
  - Exelixis Clinical Site #90, Strasbourg
  - Exelixis Clinical Site #42, Toulouse
  - Exelixis Clinical Site #67, Vandœuvre-lès-Nancy
  - Exelixis Clinical Site #37, Villejuif
- Germany (8):
  - Exelixis Clinical Site #127, Heidelberg, Baden-Wurttemberg
  - Exelixis Clinical Site #115, Tübingen, Baden-Wurttemberg
  - Exelixis Clinical Site #117, Frankfurt am Main, Hesse
  - Exelixis Clinical Site #139, Münster, North Rhine-Westphalia
  - Exelixis Clinical Site #171, Münster, North Rhine-Westphalia
  - Exelixis Clinical Site #164, Mainz, Rhineland-Palatinate
  - Exelixis Clinical Site #137, Jena, Thuringia
  - Exelixis Clinical Site #124, Dresden
- Hong Kong (3):
  - Exelixis Clinical Site #28, Hong Kong
  - Exelixis Clinical Site #136, Shatin
  - Exelixis Clinical Site #111, Tuenmen
- Hungary (2):
  - Exelixis Clinical Site #39, Budapest
  - Exelixis Clinical Site #51, Pécs
- Israel (6):
  - Exelixis Clinical Site #88, Beersheba
  - Exelixis Clinical Site #81, Haifa
  - Exelixis Clinical Site #84, Jerusalem
  - Exelixis Clinical Site #121, Kfar Saba
  - Exelixis Clinical Site #97, Petah Tikva
  - Exelixis Clincal Site #129, Ramat Gan
- Italy (8):
  - Exelixis Clinical Site #41, Meldola, Forli - Cesena
  - Exelixis Clinical Site #70, Faenza, Ravenna
  - Exelixis Clinical Site #47, Arezzo
  - Exelixis Clinical Site #60, Modena
  - Exelixis Clinical Site #61, Padua
  - Exelixis Clinical Site #59, Pavia
  - Exelixis Clinical Site #104, Perugia
  - Exelixis Clinical Site #68, Terni
- Mexico (8):
  - Exelixis Clinical Site #123, Aguascalientes, Aguascalientes
  - Exelixis Clinical Site #167, León, Guanajuato
  - Exelixis Clinical Site #169, Zapopan, Jalisco
  - Exelixis Clinical Site #134, Monterrey, Nuevo León
  - Exelixis Clinical Site #132, Oaxaca City, Oaxaca
  - Exelixis Clinical Site #160, Mexico City
  - Exelixis Clinical Site #131, Querétaro
  - Exelixis Clinical Site #161, Querétaro
- Netherlands (2):
  - Exelixis Clinical Site #144, Amsterdam
  - Exelixis Clinical Site #149, Rotterdam
- New Zealand (2):
  - Exelixis Clinical Site #122, Hamilton, Waikato Region
  - Exelixis Clinical Site #148, Newtown, Wellington Region
- Poland (5):
  - Exelixis Clinical Site #31, Biała Podlaska
  - Exelixis Clinical Site #62, Bydgoszcz
  - Exelixis Clinical Site #135, Gdansk
  - Exelixis Clinical Site #99, Otwock
  - Exelixis Clinical Site #83, Poznan
- Singapore (2):
  - Exelixis Clinical Site #77, Singapore
  - Exelixis Clinical Site #40, Singapore
- South Korea (4):
  - Exelixis Clinical Site #147, Seongnam-si, Gyeonggi-do
  - Exelixis Clinical Site #143, Seoul
  - Exelixis Clinical Site #151, Seoul
  - Exelixis Clinical Site #152, Seoul
- Spain (11):
  - Exelixis Clinical Site #53, Santiago de Compostela, Coruña
  - Exelixis Clinical Site #45, Pamplona, Navarre
  - Exelixis Clinical Site #43, Barcelona
  - Exelixis Clinical Site #36, Barcelona
  - Exelixis Clinical Site #49, Córdoba
  - Exelixis Clinical Site #34, Madrid
  - Exelixis Clinical Site #94, Madrid
  - Exelixis Clinical Site #20, Madrid
  - Exelixis Clinical Site #55, Madrid
  - Exelixis Clinical Site #96, Oviedo
  - Exelixis Clinical Site #74, Valencia
- Taiwan (3):
  - Exelixis Clinical Site #142, Taichung
  - Exelixis Clinical Site #138, Taipei
  - Exelixis Clinical Site #173, Taoyuan District
- United Kingdom (5):
  - Exelixis Clinical Site #72, Cambridge
  - Exelixis Clinical Site #93, Glasgow
  - Exelixis Clinical Site #30, London
  - Exelixis Clinical Site #172, London
  - Exelixis Clinical Site #92, Manchester

REFERENCES:
- [Derived] Choueiri TK, Powles T, Albiges L, Burotto M, Szczylik C, Zurawski B, Yanez Ruiz E, Maruzzo M, Suarez Zaizar A, Fein LE, Schutz FA, Heng DYC, Wang F, Mataveli F, Chang YL, van Kooten Losio M, Suarez C, Motzer RJ; COSMIC-313 Investigators. Cabozantinib plus Nivolumab and Ipilimumab in Renal-Cell Carcinoma. N Engl J Med. 2023 May 11;388(19):1767-1778. doi: 10.1056/NEJMoa2212851. PMID 37163623
- [Derived] Labriola MK, George DJ. Setting a new standard for long-term survival in metastatic kidney cancer. Cancer. 2022 Jun 1;128(11):2058-2060. doi: 10.1002/cncr.34177. Epub 2022 Apr 5. No abstract available. PMID 35383907
- [Derived] Mar N, Kaakour D, Rezazadeh Kalebasty A. Renal Cell Carcinoma-Lessons in Diversity, Breakthroughs, and Challenges. JCO Oncol Pract. 2022 Mar;18(3):197-199. doi: 10.1200/OP.21.00446. Epub 2021 Sep 22. No abstract available. PMID 34550754
- [Derived] Hofmann F, Hwang EC, Lam TB, Bex A, Yuan Y, Marconi LS, Ljungberg B. Targeted therapy for metastatic renal cell carcinoma. Cochrane Database Syst Rev. 2020 Oct 14;10(10):CD012796. doi: 10.1002/14651858.CD012796.pub2. PMID 33058158

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results reported in this study are based upon the data cutoff date of 09 May 2024.
Groups:
- Cabozantinib + Nivolumab + Ipilimumab: Participants received cabozantinib 40 milligrams (mg) orally once daily (qd) + 4 doses of nivolumab 3 milligrams/kilograms (mg/kg) infusion once every 3 weeks (q3w) + 4 doses of ipilimumab 1 mg/kg infusion q3w followed by cabozantinib 40 mg orally qd + nivolumab 480 mg infusion once every 4 weeks (q4w).
- Placebo + Nivolumab + Ipilimumab: Participants received cabozantinib matched placebo orally qd + 4 doses of nivolumab 3 mg/kg infusion q3w + 4 doses of ipilimumab 1 mg/kg infusion q3w followed by cabozantinib matched placebo orally qd + nivolumab 480 mg infusion q4w.
Period: Overall Study
Arm/Group | Cabozantinib + Nivolumab + Ipilimumab | Placebo + Nivolumab + Ipilimumab
Started | 428 | 427
Received at Least 1 Dose of Study Drug | 426 | 423
Progression Free Survival (PFS) Intent-to-Treat (PITT) Population (PFS Intent-to-Treat (PITT) population was defined as the first 550 randomized participants regardless of whether any study treatment or the correct study treatment was received.) | 276 | 274
Safety Analysis Set (The Safety population consisted of all participants who received any amount of study treatment.) | 426 | 423
Intent to Treat (ITT) Population (The ITT population consisted of all participants who were randomized, regardless of whether any study treatment or the correct study treatment is received.) | 428 | 427
Completed | 185 | 187
Not Completed | 243 | 240
Not completed — Death | 223 | 211
Not completed — Withdrawal by Subject | 17 | 25
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population was defined as all randomized participants regardless of whether any study treatment or the correct study treatment was received.
Groups:
- Cabozantinib + Nivolumab + Ipilimumab: Participants received cabozantinib 40 mg orally qd + 4 doses of nivolumab 3 mg/kg infusion q3w + 4 doses of ipilimumab 1 mg/kg infusion q3w followed by cabozantinib 40 mg orally qd + nivolumab 480 mg infusion q4w.
- Total: Total of all reporting groups
Arm/Group | Cabozantinib + Nivolumab + Ipilimumab | Placebo + Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 428 | 427 | 855
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 277 | 276 | 553
  >=65 years | 151 | 151 | 302
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 115 | 217
  Male | 326 | 312 | 638
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130 | 127 | 257
  Not Hispanic or Latino | 263 | 273 | 536
  Unknown or Not Reported | 35 | 27 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 10 | 14
  Asian | 29 | 33 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 3 | 6 | 9
  White | 339 | 331 | 670
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 51 | 43 | 94

OUTCOME MEASURES:

1. Primary Outcome: Duration of Progression-Free Survival (PFS) by Blinded Independent Radiology Committee (BIRC)
Description: Duration of PFS was defined as the time from randomization to the earlier of either the date of radiographic progression per BIRC or the date of death due to any cause. PFS (months) = (earliest date of progression, death, censoring - date of randomization + 1)/30.4375. PFS was determined as per Response Evaluation Criteria in Solid Tumors version (RECIST) v1.1.
Time Frame: Up to 32 months
Population: PFS Intent-to-Treat (PITT) population was defined as the first 550 randomized participants regardless of whether any study treatment or the correct study treatment was received. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib + Nivolumab + Ipilimumab | Placebo + Nivolumab + Ipilimumab
Number analyzed (Participants) | 116 | 133
months | NA [14.00 to NA] — NA signifies that the median and upper limit of 95% CI was not estimable due to a low number of events observed. | 11.30 [7.69 to 18.17]
Statistical Analysis 1: Comparison: Cabozantinib + Nivolumab + Ipilimumab vs Placebo + Nivolumab + Ipilimumab; Test type: Superiority; p = 0.0131, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.57 to 0.94]

2. Secondary Outcome: Duration of Overall Survival (OS)
Description: Duration of OS (months) = (earliest date of death or censoring - date of randomization + 1)/30.4375.
Time Frame: Up to 58 months
Population: The ITT population was defined as all randomized participants regardless of whether any study treatment or the correct study treatment was received. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib + Nivolumab + Ipilimumab | Placebo + Nivolumab + Ipilimumab
Number analyzed (Participants) | 226 | 217
months | 41.86 [34.79 to 47.87] | 41.99 [34.92 to 53.13]

ADVERSE EVENTS:
Time Frame: Day 1 up to 58 months
Description: The Safety population consisted of all participants who received any amount of study treatment. Data for All-Cause Mortality were collected for the safety analysis set.
Arm/Group | Cabozantinib + Nivolumab + Ipilimumab | Placebo + Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 224/426 | 217/423
Serious Adverse Events (participants affected / at risk) | 272/426 | 257/423
Other Adverse Events (participants affected / at risk) | 421/426 | 416/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib + Nivolumab + Ipilimumab (N=426) | Placebo + Nivolumab + Ipilimumab (N=423)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acquired factor VIII deficiency (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 6 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 6
Myocarditis (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 0 | 2
Autoimmune myocarditis (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 11 | 12
Hypophysitis (Endocrine disorders) | 2 | 7
Hyperthyroidism (Endocrine disorders) | 3 | 2
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 1 | 0
Immune-mediated thyroiditis (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 1 | 0
Orbital myositis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 17
Colitis (Gastrointestinal disorders) | 5 | 10
Vomiting (Gastrointestinal disorders) | 2 | 9
Nausea (Gastrointestinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 6
Intestinal obstruction (Gastrointestinal disorders) | 2 | 3
Ascites (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Malabsorption (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Overflow diarrhoea (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 4
General physical health deterioration (General disorders) | 5 | 6
Asthenia (General disorders) | 3 | 3
Death (General disorders) | 2 | 4
Fatigue (General disorders) | 3 | 2
Disease progression (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 2
Sudden death (General disorders) | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 2
Multiple organ dysfunction syndrome (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Condition aggravated (General disorders) | 0 | 1
Crepitations (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
Swelling face (General disorders) | 1 | 0
Ulcer (General disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 20 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 7 | 4
Hepatitis (Hepatobiliary disorders) | 5 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 16 | 17
Pneumonia (Infections and infestations) | 13 | 10
Sepsis (Infections and infestations) | 6 | 5
Anal abscess (Infections and infestations) | 5 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 2 | 2
Diverticulitis (Infections and infestations) | 1 | 2
Empyema (Infections and infestations) | 2 | 1
Meningitis aseptic (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Appendicitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Human anaplasmosis (Infections and infestations) | 0 | 1
Infected fistula (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Sciatic nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 45 | 11
Aspartate aminotransferase increased (Investigations) | 34 | 13
Lipase increased (Investigations) | 6 | 1
Blood bilirubin increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 3 | 1
Amylase increased (Investigations) | 3 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 2 | 1
Transaminases increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Haemoglobin increased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 0 | 1
Troponin T increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Cell death (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 7
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 15
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 8
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seizure (Nervous system disorders) | 1 | 4
Cerebrovascular accident (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Brain oedema (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cervical cord compression (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Embolic cerebellar infarction (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Immune-mediated encephalitis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 4
Haematuria (Renal and urinary disorders) | 3 | 6
Renal failure (Renal and urinary disorders) | 2 | 4
Nephritis (Renal and urinary disorders) | 1 | 4
Immune-mediated nephritis (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Autoimmune nephritis (Renal and urinary disorders) | 0 | 1
Bladder hypertrophy (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Paraphimosis (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal mucosa atrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 7 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Cyanosis (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib + Nivolumab + Ipilimumab (N=426) | Placebo + Nivolumab + Ipilimumab (N=423)
Anaemia (Blood and lymphatic system disorders) | 77 | 94
Neutropenia (Blood and lymphatic system disorders) | 29 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 6
Hypothyroidism (Endocrine disorders) | 122 | 81
Hyperthyroidism (Endocrine disorders) | 54 | 48
Diarrhoea (Gastrointestinal disorders) | 216 | 108
Nausea (Gastrointestinal disorders) | 112 | 105
Vomiting (Gastrointestinal disorders) | 78 | 66
Constipation (Gastrointestinal disorders) | 64 | 66
Abdominal pain (Gastrointestinal disorders) | 72 | 41
Stomatitis (Gastrointestinal disorders) | 68 | 11
Dry mouth (Gastrointestinal disorders) | 38 | 40
Dyspepsia (Gastrointestinal disorders) | 44 | 23
Abdominal pain upper (Gastrointestinal disorders) | 28 | 25
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 29 | 12
Fatigue (General disorders) | 133 | 129
Asthenia (General disorders) | 103 | 68
Pyrexia (General disorders) | 78 | 61
Oedema peripheral (General disorders) | 43 | 36
Mucosal inflammation (General disorders) | 50 | 17
Chest pain (General disorders) | 16 | 25
Hypertransaminasaemia (Hepatobiliary disorders) | 24 | 10
COVID-19 (Infections and infestations) | 62 | 52
Urinary tract infection (Infections and infestations) | 42 | 34
Alanine aminotransferase increased (Investigations) | 204 | 89
Aspartate aminotransferase increased (Investigations) | 195 | 74
Lipase increased (Investigations) | 106 | 78
Amylase increased (Investigations) | 100 | 66
Blood creatinine increased (Investigations) | 68 | 62
Weight decreased (Investigations) | 50 | 39
Gamma-glutamyltransferase increased (Investigations) | 45 | 31
Blood bilirubin increased (Investigations) | 45 | 18
Blood alkaline phosphatase increased (Investigations) | 42 | 16
Blood thyroid stimulating hormone increased (Investigations) | 28 | 17
Blood lactate dehydrogenase increased (Investigations) | 22 | 9
Decreased appetite (Metabolism and nutrition disorders) | 118 | 84
Hyponatraemia (Metabolism and nutrition disorders) | 48 | 42
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 32
Hypomagnesaemia (Metabolism and nutrition disorders) | 40 | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 22 | 21
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 16
Hypophosphataemia (Metabolism and nutrition disorders) | 27 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 25 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 96 | 96
Back pain (Musculoskeletal and connective tissue disorders) | 62 | 68
Pain in extremity (Musculoskeletal and connective tissue disorders) | 46 | 39
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 47 | 9
Headache (Nervous system disorders) | 70 | 65
Dizziness (Nervous system disorders) | 38 | 38
Dysgeusia (Nervous system disorders) | 45 | 16
Insomnia (Psychiatric disorders) | 43 | 34
Proteinuria (Renal and urinary disorders) | 42 | 43
Haematuria (Renal and urinary disorders) | 30 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 66 | 62
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 41
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 61 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 106 | 131
Rash (Skin and subcutaneous tissue disorders) | 105 | 97
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 123 | 26
Dry skin (Skin and subcutaneous tissue disorders) | 31 | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 28 | 17
Hypertension (Vascular disorders) | 125 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03937219/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03937219/SAP_001.pdf